CLINICAL TRIAL: NCT07070947
Title: Efficacy of Manual Therapy in Indirect Non-Invasive Neuromodulation of the Vagus Nerve in the Treatment of Bruxism in Young Adult Population up to 40 Years Old
Brief Title: Surface Electromyography in the Detection and Assessment of Bruxism
Acronym: EMGBruxism
Status: Not yet recruiting | Type: Observational
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Maider Sánchez Padilla, MSc, Escoles Universitaries Gimbernat
Other Study IDs: EMGBruxism
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Bruxism, Sleep
Keywords: Sleep Bruxism; Electromyography; Masticatory Muscles
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Bruxism): Temporomandibular disorder: Active symptoms compatible with nocturnal bruxism according to ICSD-III and RDC/TMD criteria
  Interventions: Diagnostic Test: sEMG
- Group 2 (No bruxism): Asymptomatic and without signs of bruxism or other craniofacial pathologies
  Interventions: Diagnostic Test: sEMG

INTERVENTIONS:
Diagnostic Test: sEMG — The spectral characteristics in the amplitude domain will be recorded through the root mean square (RMS, unit: μV) or the mean power frequency (MPF, unit: Hz) of the musculature to be evaluated by means of EMGs, with the electrodes placed parallel to the muscle fibers of the temporal, masseter, and suprahyoid muscles. Standardized EMGs will be recorded and compared in resting position and during maximum voluntary clenching

SUMMARY:
Introduction:

Sleep bruxism is defined as the repetitive activity of the masticatory muscles, characterized by clenching or grinding of the teeth. Studies confirm the association between sleep bruxism and episodes of masticatory muscle activity, with an increase in autonomic sympathetic activity observed during transient periods of sleep. This is associated with nocturnal awakenings, related to increased cardiac, cerebral (cortical arousal), respiratory, and muscular activity.

Objectives: The main objectives are "To study the mean power frequency (MPF) of the masticatory muscles measured by surface electromyography (sEMG) in the general population (with and without bruxism according to ICSD-3 and DC/TMD criteria)"; and "to assess the effectiveness of manual therapy applied to structures adjacent to the vagus nerve based on its impact on orofacial pain and symptomatology in patients with bruxism".

Material and Methods:

A cross-sectional observational study and a randomized controlled experimental study were designed. The first will analyze data collected by sEMG in the masticatory muscles, at rest and during maximum clenching, comparing results between bruxists and non-bruxists. The second will analyze, compared to the control group, data collected on signs (range of motion alteration, presence of sounds), symptomatology (pain, headaches, sensation of blockage, functional limitation) caused by bruxism, sleep quality (Pittsburgh Sleep Quality Index (PSQI)), oral health-related quality of life (OHIP-14), stress and anxiety status (Perceived Stress Scale and GAD-7 (Generalized Anxiety Disorder-7), respectively), and sympathetic-vagal balance (Heart Rate Variability in its frequency and time domains) before and after a manual therapy intervention on structures adjacent to the vagus nerve pathway (head, neck, thorax, diaphragm, abdomen). The collected data will be analyzed using IBM SPSS® version 25.0.0.

ELIGIBILITY:
Inclusion Criteria:

For patients with bruxism:

1. Sleep bruxism diagnosed according to the ICSD-III (International Classification of Sleep Disorders, 3rd edition):

   * Regular or frequent tooth grinding sounds occurring during sleep and the presence of one or more of the following clinical signs and symptoms:

     1. Abnormal tooth wear consistent with reports of clenching/grinding the teeth during sleep
     2. Transient morning pain or fatigue in the jaw muscles; and/or temporal headaches; and/or jaw locking upon awakening, consistent with reports of clenching/grinding the teeth during sleep
2. Sleep bruxism diagnosed according to the RDC/TMD:

   * Interview: During the interview, subjects are asked about the following symptoms: reports of regular or frequent tooth grinding during sleep, muscle fatigue, temporal headache, transient morning muscle pain in the jaw, and jaw locking upon awakening.
   * Physical examination: Presence or signs suggesting abnormal dental wear, such as teeth with flattened cusps and/or loss of contour with dentin exposure.

     * Hypertrophy of the masticatory muscles
     * Dental impressions on the tongue
     * Linea alba on the cheeks along the bite line
     * Damage to dental tissue
     * Excessive dental wear
3. A minimum pain intensity score of 3 on the Visual Analogue Scale at the masseter and temporal algometry points.
4. EMGs with elevated mean power frequency for the masseter and temporalis muscles (to be defined in the first clinical phase-observational study).
5. Age between 18 and 40 years.

For patiens without bruxism:

a)Asymptomatic and without signs of bruxism or other craniofacial pathologies.

Exclusion Criteria:

1. Having suffered direct trauma, mandibular fractures, or surgeries in the orofacial region.
2. Loss of more than 2 teeth, except for the third molar.
3. Use of muscle relaxant medication or medications that may influence motor behavior.
4. Having received botulinum toxin treatment in the last 6 months.
5. Periodontal disorders or current orthodontic treatment or prosthesis.
6. Partial or total dentures.
7. History of medical disorders (severe psychiatric, physiological, or neurological conditions).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The observational study will include two groups of patients: the first, with active symptoms compatible with nocturnal bruxism, and the second, asymptomatic patients without signs of bruxism or other craniofacial pathologies. To this end, 54 participants aged between 18 and 40 years will be recruited.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor recruitment pattern of the masseter, temporalis, and suprahyoid muscles | 1 day, baseline
  In resting position and during maximum clenching, as measured by the mean power frequency (MPF) recorded in a surface electromyography.

SECONDARY OUTCOMES:
Orofacial Pain (1) | 1 day, baseline
  Assessment tests for TMD and bruxism condition "AXIS- I" is the assessment tool with a "Symptom questionnaire"
Orofacial Pain (2) | 1 day, baseline
  Assessment tests for TMD and bruxism condition "AXIS- I" is the assessment tool with a Pressure Pain Threshold of masseter and temporalis muscles with a DC/ TMD EXAMINATION FORM.
Orofacial Pain (3) | 1 day, baseline
  Assessment tests for TMD and bruxism condition "AXIS -II" throught the "Graded chronic pain scale version 2.0"
Range of Motion (1) | 1 day, baseline
  Assessment tests for TMD and bruxism condition "AXIS- I" is the assessment tool with a "Symptom questionnaire".
Range of Motion (2) | 1 day, baseline
  Assessment tests for TMD and bruxism condition "AXIS- I" is the assessment tool with a range of motion with a DC/ TMD EXAMINATION FORM.
Jaw Funcionality | 1 day, baseline
  AXIS-II" is the assesment tool that include "Jaw Functional Limitation Scale-20
Oral behavior | 1 day, baseline
  AXIS-II" is the assesment tool that include "The Oral Behavior checklist
Headaches | 1 day, baseline
  The assessment will be carried out using HIT-6 (Headeach Impact Test-6)
Sleep Quality | 1 day, baseline
  Sleep quality is considered one of the most important measures related to bruxism. To assess it, the Pittsburgh Sleep Quality Index (PSQI) questionnaire will be administered.
Oral health-related quality of life | 1 day, baseline
  To assess it, the HIP-14 (Oral Health Impact Profile-14) questionnaire will be administered.
Stress | 1 day, baseline
  To assess it, the PPS: Perceived Stress Scale will be administered.
Anxiety | 1 day, baseline
  To assess it, the GAD-7 (General Anxiety Disorder-7) will be administered.
Heart Rate Variability (HRV) | 1 day, baseline
  Spectral analysis of the time variation between consecutive heartbeats, referred to as the RR interval, which records the activity of the autonomic nervous system. This is collected using the chest strap "Polar H10 Band," which connects to the mobile app "Elite HRV" or "Kubios Software." It collects the frequency measures: LF (low frequency), HF (high frequency), and the ratio between them (LF/HF) as an indicator of sympathetic-vagal balance. It collects the time-domain measures: Mean RR interval; SDNN: standard deviation of all RR intervals; pNN50; RMSSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat International de Catalunya (UIC), Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Once the project is completed, the all IPD collected throughout the trial will be disseminated through presentations at various national and international conferences.
  Manuscripts describing the IPD collected will also be prepared and submitted for publication in peer-reviewed journals.

REFERENCES:
- [Background] Abe S, Huynh NT, Kato T, Rompre PH, Landry-Schonbeck A, Landry ML, de Grandmont P, Kawano F, Lavigne GJ. Oral appliances reduce masticatory muscle activity-sleep bruxism metrics independently of changes in heart rate variability. Clin Oral Investig. 2022 Sep;26(9):5653-5662. doi: 10.1007/s00784-022-04520-y. Epub 2022 May 10. PMID 35538329
- [Background] Matusz K, Maciejewska-Szaniec Z, Gredes T, Pobudek-Radzikowska M, Glapinski M, Gorna N, Przystanska A. Common therapeutic approaches in sleep and awake bruxism - an overview. Neurol Neurochir Pol. 2022;56(6):455-463. doi: 10.5603/PJNNS.a2022.0073. Epub 2022 Nov 29. PMID 36444852
- [Background] Amorim CSM, Espirito Santo AS, Sommer M, Marques AP. Effect of Physical Therapy in Bruxism Treatment: A Systematic Review. J Manipulative Physiol Ther. 2018 Jun;41(5):389-404. doi: 10.1016/j.jmpt.2017.10.014. PMID 30041736
- [Background] Kuang B, Li D, Lobbezoo F, de Vries R, Hilgevoord A, de Vries N, Huynh N, Lavigne G, Aarab G. Associations between sleep bruxism and other sleep-related disorders in adults: a systematic review. Sleep Med. 2022 Jan;89:31-47. doi: 10.1016/j.sleep.2021.11.008. Epub 2021 Nov 19. PMID 34879286
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Thymi M, Shimada A, Lobbezoo F, Svensson P. Clinical jaw-muscle symptoms in a group of probable sleep bruxers. J Dent. 2019 Jun;85:81-87. doi: 10.1016/j.jdent.2019.05.016. Epub 2019 May 11. PMID 31085350
- [Background] Michalek-Zrabkowska M, Martynowicz H, Wieckiewicz M, Smardz J, Poreba R, Mazur G. Cardiovascular Implications of Sleep Bruxism-A Systematic Review with Narrative Summary and Future Perspectives. J Clin Med. 2021 May 21;10(11):2245. doi: 10.3390/jcm10112245. PMID 34064229
- [Background] Schaffarczyk M, Rogers B, Reer R, Gronwald T. Validity of the Polar H10 Sensor for Heart Rate Variability Analysis during Resting State and Incremental Exercise in Recreational Men and Women. Sensors (Basel). 2022 Aug 30;22(17):6536. doi: 10.3390/s22176536. PMID 36081005
- [Background] Perrotta AS, Jeklin AT, Hives BA, Meanwell LE, Warburton DER. Validity of the Elite HRV Smartphone Application for Examining Heart Rate Variability in a Field-Based Setting. J Strength Cond Res. 2017 Aug;31(8):2296-2302. doi: 10.1519/JSC.0000000000001841. PMID 28195974
- [Background] Matusik PS, Zhong C, Matusik PT, Alomar O, Stein PK. Neuroimaging Studies of the Neural Correlates of Heart Rate Variability: A Systematic Review. J Clin Med. 2023 Jan 28;12(3):1016. doi: 10.3390/jcm12031016. PMID 36769662
- [Background] von Piekartz H, Bleiss S, Herzer S, Hall T, Ballenberger N. Does combining oro-facial manual therapy with bruxism neuroscience education affect pain and function in cases of awake bruxism? A pilot study. J Oral Rehabil. 2024 Sep;51(9):1692-1700. doi: 10.1111/joor.13740. Epub 2024 Jun 18. PMID 38894567
- [Background] Wojcik M, Siatkowski I. The effect of cranial techniques on the heart rate variability response to psychological stress test in firefighter cadets. Sci Rep. 2023 May 13;13(1):7780. doi: 10.1038/s41598-023-34093-z. PMID 37179419
- [Background] Kadioglu MB, Sezer M, Elbasan B. Effects of Manual Therapy and Home Exercise Treatment on Pain, Stress, Sleep, and Life Quality in Patients with Bruxism: A Randomized Clinical Trial. Medicina (Kaunas). 2024 Dec 4;60(12):2007. doi: 10.3390/medicina60122007. PMID 39768887
- [Background] Berni KC, Dibai-Filho AV, Pires PF, Rodrigues-Bigaton D. Accuracy of the surface electromyography RMS processing for the diagnosis of myogenous temporomandibular disorder. J Electromyogr Kinesiol. 2015 Aug;25(4):596-602. doi: 10.1016/j.jelekin.2015.05.004. Epub 2015 May 27. PMID 26054969
- [Background] Lodetti G, Mapelli A, Musto F, Rosati R, Sforza C. EMG spectral characteristics of masticatory muscles and upper trapezius during maximum voluntary teeth clenching. J Electromyogr Kinesiol. 2012 Feb;22(1):103-9. doi: 10.1016/j.jelekin.2011.10.008. Epub 2011 Nov 17. PMID 22100151
- [Background] Lobbezoo F, Aarab G, Ahlers MO, Baad-Hansen L, Bernhardt O, Castrillon EE, Giannakopoulos NN, Gronbeck A, Hauschild J, Holst-Knudsen M, Skovlund N, Thymi M, Svensson P. Consensus-based clinical guidelines for ambulatory electromyography and contingent electrical stimulation in sleep bruxism. J Oral Rehabil. 2020 Feb;47(2):164-169. doi: 10.1111/joor.12876. Epub 2019 Sep 11. PMID 31430389
- [Background] Merletti R, Muceli S. Tutorial. Surface EMG detection in space and time: Best practices. J Electromyogr Kinesiol. 2019 Dec;49:102363. doi: 10.1016/j.jelekin.2019.102363. Epub 2019 Oct 19. PMID 31665683
- [Background] Nalamliang N, Sumonsiri P, Thongudomporn U. Masticatory performance is influenced by masticatory muscle activity balance and the cumulative occlusal contact area. Arch Oral Biol. 2021 Jun;126:105113. doi: 10.1016/j.archoralbio.2021.105113. Epub 2021 Mar 30. PMID 33826961